CLINICAL TRIAL: NCT06409962
Title: A New Technological Intervention to Address Childhood Obesity: Approach to Multidimensional Intervention
Brief Title: A New Technological Intervention to Address Childhood Obesity:
Acronym: NURSPEDIAOBE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Córdoba (Other)
Collaborators: Instituto Maimónides de Investigación Biomédica de Córdoba (IMIBIC) (Unknown)
Responsible Party: Principal Investigator, Pilar Aparicio Martinez, Assistant Professor, Universidad de Córdoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5345
Record Dates: First submitted 2024-04-17; First posted 2024-05-10 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Body Weight; Dyslipidemias; Musculoskeletal Diseases
Keywords: pediatric; body mass index; intervention; anthopometric; blood pressure
MeSH Terms: conditions — Body Weight; Dyslipidemias; Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: Our proposed intervention, which integrates nutritional intervention with the use of innovative technologies, holds significant potential for yielding tangible outcomes in the prevention and management of this condition within the region. By doing so, it mitigates the risk of overweight and obesity-related pathologies in adulthood.
  The inclusion of both experimental and control groups in the sample distribution will facilitate an effective evaluation of the nutritional intervention, offering concrete data on the efficacy of the implemented strategies. Furthermore, the comprehensive assessment encompassing anthropometric measurements, biometric data, and physical activity records will provide a detailed understanding of the intervention's effects on the school population.
Who Masked: Investigator
Masking Description: The randomisation will be conducted based on an artificial model, utilising a coding system that assigns numerical identifiers to names, postal codes, and grade levels. This approach ensures a systematic and unbiased selection process, allowing for a fair representation of participants across various demographic factors.
  The sampling has been estimaited by Epidat program. The experimental group, receiving nutritional intervention, will consist of approximately 50% of the total sample, equivalent to 215 participants. Meanwhile, the control group, not receiving the intervention, will comprise the remaining 50% of the sample, also around 215 participants. This distribution will enable an effective comparison of results between the two groups and assess the effectiveness of the nutritional intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Technological intervention (Experimental): The experimental arm integrates technology-based interventions-podcasts, gamification, and virtual reality-to promote nutritional education and healthy behaviors. Tailored podcasts cover topics like healthy eating habits and balanced nutrition, while gamification enhances motivation. Virtual reality offers immersive environments for exploring healthy choices. Both experimental and control groups enable a comprehensive evaluation, collecting data through measurements, biometrics, and activity records.
  Interventions: Other: Technological combination
- No-technological intervention: traditional brochure (No Intervention): The control arm will focus on a non-technological intervention, specifically utilizing traditional brochures. Participants in this arm will receive printed materials containing information on basic nutritional guidelines, healthy eating habits, and the importance of balanced nutrition. The brochure-based intervention aims to provide essential information in a straightforward format, emphasizing key messages related to healthy eating practices. Participants will have access to pamphlets outlining dietary recommendations, portion control, and tips for making nutritious food choices.

INTERVENTIONS:
Other: Technological combination — The intervention comprises workshops, individualized counseling, cooking classes, and physical activity promotion. It emphasizes nutritional education, hands-on cooking, and behavioral modification techniques. Participants receive personalized guidance and resources to make sustainable dietary and lifestyle changes. Social support networks foster motivation and accountability. By combining these components, the intervention aims to empower participants with the knowledge, skills, and support needed for long-term health improvements.
  Other Names: Impact of technology on healthy lifestyle
  Arms: Technological intervention

SUMMARY:
Childhood obesity is a global public health issue, with rising prevalence rates. In Spain, the problem is significant, particularly in the southern regions. Factors contributing to childhood obesity include dietary habits, lack of physical activity, and socioeconomic influences.

Efforts to address childhood obesity in Spain include various programs focusing on dietary modification, increased physical activity, and family involvement. Despite these initiatives, there is a need for continued intervention, as changing dietary and lifestyle patterns have led to reduced fruit and vegetable consumption and increased sedentary behavior among children.

Childhood obesity has concerning health implications, including heart-related issues. Echocardiography plays a vital role in early detection.

Given the limited research on the impact of childhood obesity on musculoskeletal development and mobility, a comprehensive study is needed to analyze its prevalence and associated factors. The study aims to assess the effectiveness of nutritional interventions administered by school nurses.

In summary, childhood obesity in Spain is a growing concern, with multifaceted causes and health implications. Ongoing efforts are required to combat this issue and promote healthier lifestyles among children.

DETAILED DESCRIPTION:
An elevated Body Mass Index (BMI) in the child population represents a significant global public health concern. According to the World Health Organization (WHO), overweight occurs in children aged 6-19 when the BMI exceeds one or more standard deviations from the median established in WHO child growth patterns.

Epidemiological data reflects that since the late 20th century, childhood obesity has increased from 4.9% (31.5 million) to 6% (40.6 million) worldwide. According to data from the Childhood Obesity Surveillance Initiative (COSI) within the European Union (EU), children in Spain aged 6-9 have a 42% overweight rate and a 19% obesity rate. In comparison, girls have a 41% overweight rate and a 17% obesity rate, positioning Spain as the fourth EU country with the highest prevalence of overweight and obesity in children.

Within the national territory, 4 out of 10 schoolchildren have excess weight, with the highest prevalence in the southern regions. The autonomous community with the lowest incidence of childhood overweight is Navarra, with 15%, and the highest is the Region of Murcia, with 40%. Andalusians present a high prevalence rate of 33.4%. In general, the country's northern regions have lower figures, while the southern region has the highest rates of childhood overweight. It has also been observed that there is a higher likelihood of being overweight in rural areas than in urban areas.

This could be due to regional differences in habits during the three critical periods for the development of childhood obesity: the preconception period involving maternal factors, the first 1000 days of life (9 months of pregnancy + 2 years of life), and the adiposity rebound between 5-7 years. Childhood overweight is also highly influenced by factors such as maternal overweight, early introduction of complementary feeding before 6 months of age, smoking during pregnancy, low parental educational levels, and the excessive use of screens such as mobile phones or tablets at an early age.

The most relevant factors in overweight are diet, physical inactivity, physical activity, and lifestyle habits. However, when it comes to minors, all these factors are strongly influenced by the cultural, social, and institutional environment, as well as the family's socioeconomic level.

In Spain, Andalusia is one of the autonomous communities with a lower income index (0.67) and a lower average expenditure on public health at 0.33%. However, the community puts in the most effort to implement policies against obesity, with a score of 5.19.

Numerous campaigns have been launched to prevent childhood obesity, developed by the Spanish Agency for Consumer Affairs, Food Safety, and Nutrition (AECOSAN) as part of the nutrition, physical activity, and obesity prevention (NAOS) strategy. Additionally, the Andalusian Ministry of Health and Families has implemented plans such as "Growing in Health," "Evaluation of Food Offer in Andalusian Schools 2019-2020," and the "Health throughout Life" campaign.

All these programs coincide on three fundamental aspects when addressing childhood obesity: interventions to modify dietary habits promoting balanced and healthy eating, increasing fruit and vegetable consumption while minimizing sugar intake; interventions to promote physical activity, encouraging at least one hour of exercise daily; and, lastly, family involvement interventions to achieve proper adherence to these changes.

These interventions are necessary today because, over the past decades, there have been changes in eating patterns and diets, resulting in a decrease in the consumption of fruits, vegetables, legumes, and fresh products, as well as an increase in the consumption of processed foods with higher sugar, fat, salt content, and poorer nutritional quality. According to COSI initiative data, Spain is where children consume the least fruits and vegetables daily. There have also been changes in physical activity, with studies showing that 25% of Spanish children are sedentary.

One of the direct consequences of childhood overweight is morphological heart alterations, reflected in left ventricular hypertrophy and cardiac diastolic alterations. Numerous scientific studies have established a close relationship between obesity in children and adolescents and an increase in epicardial fat, which can lead to cardiac and vascular abnormalities. In fact, having a high BMI at a young age has become a significant risk factor for the premature development of cardiovascular diseases that were previously considered exclusive to adults. These changes are visible through echocardiography, especially in epicardial fat.

As a non-invasive diagnostic tool, Echocardiography has gained a fundamental role in early detection of these alterations in the pediatric population affected by an increase in epicardial fat. Its early implementation allows for precise cardiac and vascular function assessment, improving these young patients' quality of life and prognosis. These measurements and modifications have been analyzed recently, although more data on younger populations and post-pandemic needs to be collected. Furthermore, to address this growing challenge, it is crucial to raise awareness about the importance of maintaining a healthy weight early and promote research and the application of preventive and intervention strategies to reduce epicardial fat in the pediatric population.

Due to all the aforementioned reasons, coupled with the limited number of current publications that deeply analyze the consequences of childhood obesity on the development of the musculoskeletal system and children's mobility, it is essential to conduct a study of the population and subsequently intervene to promote healthy growth and development in children.

Therefore, the objective is to establish the impact of a nutritional intervention by a school nurse on a group of schoolchildren.

ELIGIBILITY:
Inclusion Criteria:

* Students from the school
* Pediatric from age 6 to 16
* Students from the school that confirmed approval
* Signed informed consent by the minor
* Signed informed consent by the minor's parents or guardians.

Exclusion Criteria:

* Presence of HbA1c levels below 5.7%
* Presence of HbA1c levels above 6.4%
* Presence of pathological metabolic diseases, such as diabetes or metabolic syndrome
* Presence of other diseases related to intestinal integrity or skin issues.
* Lack of the signed informed consent by the minor and legal guardian

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 215 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2026-12-12 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight (kg) | From 12 weeks (1st measurement) up 15th months (6th measurement)
  Weight, as a pivotal anthropometric measure, will be quantified using a validated weight machine, alongside a body composition monitor such as the BF511. The validated weight machine adheres to established calibration standards, ensuring precision and consistency in measurements. It employs advanced technology to accurately assess an individual's weight in kilograms (kg), providing reliable data for scientific analyses.
Height (m2) | From 12 weeks (1st measurement) up 15th months (6th measurement)
  Height will be registered in meters squared (m^2) for its precise evaluation. Employing a validated tachymeter, a specialized instrument designed for accurate measurements, ensures meticulous assessment of height.
Percentage Lean Mass (LM) (%) | From 12 weeks (1st measurement) up 15th months (6th measurement)
  The lean fat, calculated in percentage, will be obtained using a validated weight machine, alongside a body composition monitor such as the BF511.
Percentage Fat Mass (FM) (%) | 1st month, 3 month, 6 month, 9 month, 12th and 15th month
  The lean fat, calculated in percentage, will be obtained using a validated weight machine, alongside a body composition monitor such as the BF511.
Body Mass Index (kg/m2) | From 12 weeks (1st measurement) up 15th months (6th measurement)
  The Body Mass Index will be calculated using the percentiles according to age group and sex.
Waist circumference (cm) | From 12 weeks (1st measurement) up 15th months (6th measurement)
  The waist circumference (cm) of the children will be measured via an inextensible measuring tape at the initial visit (1st month or V0) and at the last visit (15th month or V6).The measurement follows the recommendations of the International Standards for Anthropometric Assessment
Hip circumference(cm) | From 12 weeks (1st measurement) up 15th months (6th measurement)
  The Hip circumference(cm) of the children will be measured via an inextensible measuring tape at the initial visit (1st month or V0) and at the last visit (15th month or V6).The measurement follows the recommendations of the International Standards for Anthropometric Assessment
Arm circumference (cm) | From 12 weeks (1st measurement) up 15th months (6th measurement)
  The arm circumference (cm) of the children will be measured via an inextensible measuring tape at the initial visit (1st month or V0) and at the last visit (15th month or V6).The measurement follows the recommendations of the International Standards for Anthropometric Assessment
Calf circumference (cm) | From 12 weeks (1st measurement) up 15th months (6th measurement)
  The arm circumference (cm) of the children will be measured via an inextensible measuring tape at the initial visit (1st month or V0) and at the last visit (15th month or V6).The measurement follows the recommendations of the International Standards for Anthropometric Assessment
Validated nutritional assessment questionnaire: adherence to the Mediterranean diet (KIDMED) | From 12 weeks (1st measurement) up 15th months (6th measurement)
  he KIDMED will be used to determine adherence to the change in diet from the initial visit (V0) and the final visit (V6). This questionnaire is formed by 16 questions related to adherence to the Mediterranean diet, in addition to 7 items complementary to the test. All questions were answered positively or negatively. Of the 16 main questions, questions number 6, 11, 14, and 16, in their affirmative answers had a negative meaning, so they were worth (-1), on the other hand, the remaining questions whose affirmative answers represented a positive value concerning the Mediterranean diet were scored with (+1). Negative responses do not score (0). According to the test, the results are grouped into different levels of adherence to the Mediterranean diet, low (score 0 to 3), medium (score 4-7), and high (8 to 12).
Food Consumption Frequency | From 12 weeks (1st measurement) up 15th months (6th measurement)
  Food Frequency Questionnaire (FFQ) will be used to determine the consumption of food and the change in diet from the initial visit (V0) and the final visit (V6). Energy and nutrient intakes were calculated using Spanish food composition tables
  Food consumption frequency refers to the rate at which individuals consume different types of food within a specific time frame, typically measured over a day, week, or month. This variable captures the frequency with which individuals consume various food groups, such as fruits, vegetables, grains, proteins, and processed foods. It provides insight into dietary patterns and habits, indicating how often individuals incorporate different foods into their regular eating routines.
Blood pressure | From 12 weeks (1st measurement) up 15th months (6th measurement)
  The systolic and diastolic blood pressure will be taken using an Omron-validated tensiometer with two measurements between 15 minutes each measurement from the 1st visit (v0) to the last (v6).

SECONDARY OUTCOMES:
3D avatar system for anthropometric measures | From 12 weeks (1st measurement) up 15th months (6th measurement)
  The validation of avatar systems based on artificial vision involves assessing the accuracy, reliability, and effectiveness of virtual representations controlled by artificial intelligence algorithms. These avatars, generated using artificial vision technology, mimic human-like behavior and interactions within virtual environments. Validation encompasses rigorous testing to ensure that avatars accurately interpret and respond to visual inputs, such as facial expressions or gestures, in a manner consistent with human perception.
  The validation of avatar systems based on artificial vision involves assessing the accuracy, reliability, and effectiveness of virtual representations controlled by artificial intelligence algorithms. The results of the model will provide, using the height and weight previously measured with the Body Composition validated weight scale, will be obtained the arm, waist, calf and arm circumferences.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Vaquero Abellan, MD, Msc, PhD, Study Director — Universidad de Córdoba; Manuel Vaquero Alvárez, MD, Msc, PhD, Principal Investigator — Maimónides Biomedical Research Institute of Córdoba; Isabel Blancas Sanchez, MD, Msc, PhD, Principal Investigator — Primary Care, Jaen
Locations (1):
- Colegio Virgen del Carmen, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: No
The data of the participants will be made available to other researchers under consideration and analysis of the research committee.

REFERENCES:
- [Result] Blancas-Sanchez IM, Del Rosal Jurado M, Aparicio-Martinez P, Quintana Navarro G, Vaquero-Abellan M, Castro Jimenez RA, Fonseca Pozo FJ. A Mediterranean-Diet-Based Nutritional Intervention for Children with Prediabetes in a Rural Town: A Pilot Randomized Controlled Trial. Nutrients. 2022 Sep 1;14(17):3614. doi: 10.3390/nu14173614. PMID 36079871